CLINICAL TRIAL: NCT05947058
Title: Multicenter Randomized Controlled Trial Comparing Hip Arthroplasty to Internal Fixation for Minimally Displaced Femoral Neck Fractures: A Pilot Study
Brief Title: Minimally Displaced Femoral Neck Fracture Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Orthopaedic Trauma Association (Other); McMaster University (Other); University of Southern California (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mark Gage, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00100917
Record Dates: First submitted 2023-06-02; First posted 2023-07-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Femoral Neck Fractures
Keywords: Minimally Displaced Femoral Neck Fractures; Arthroplasty; Internal Fixation
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroplasty (Experimental): A modern porous-coated press-fit or cemented hip arthroplasty prosthesis will be used at the treating surgeon's discretion. Press-fit implants that have no ingrowth or ongrowth surface will not be permitted. We recommend surgeons consider a total hip arthroplasty for younger active, independent participants; conversely, a hemiarthroplasty is recommended for more frail, lower-demand participants. Similarly, cemented arthroplasty for older adult participants is also recommended. The surgical approach and the use of post-operative hip precautions will be determined by the treating surgeon.
  Interventions: Procedure: Arthroplasty
- Internal Fixation (Active Comparator): Based on the fracture displacement eligibility criteria, minimal or no reduction is expected during the surgical procedure. However, the treating surgeon will be allowed to perform fracture reduction maneuvers if desired. Fixed angle devices and multiple screws will be permitted. The internal fixation device(s) will be inserted through a small lateral incision. If using multiple cancellous screws, an inverted triangle or similar screw pattern is recommended. Fixed angle devices, such as a sliding hip screw (with or without an anti-rotation screw) or newer multi-screw fixed angle devices will also be permitted. Internal fixation constructs combining cancellous screws and fixed angle devices will be permitted.
  Interventions: Procedure: Internal Fixation

INTERVENTIONS:
Procedure: Arthroplasty — The type of hip prothesis (hemi or total; cemented or uncemented) will be at the discretion of the treating surgeon.
  Arms: Arthroplasty
Procedure: Internal Fixation — Both fixed angle devices and multiple screws will be permitted for the internal fixation group.
  Arms: Internal Fixation

SUMMARY:
The goal of this randomized pilot study is to assess feasibility of the trial and to collect information to inform the design of a definitive trial. Adult patients ages 60 years or older with a low-energy minimally displaced femoral neck fracture (FNF) treated with surgery will be eligible to participate in the study. Patients will be randomized to one of two treatment groups, hip arthroplasty or internal fixation. Participants will be followed for 1 year.

DETAILED DESCRIPTION:
Nearly half of all elderly hip fractures are femoral neck fractures (FNFs) and approximately 20% are minimally displaced. Internal fixation has remained the treatment of choice for these injuries because these fractures can be fixed in situ and the surgical implants can be inserted with little surgical dissection. Patients treated with internal fixation experience high complication rates, with the pooled risk of reoperation and mortality each above 14%. Preliminary data have suggested arthroplasty for minimally displaced fractures may lead to better patient outcomes, including improved ambulation, fewer reoperations, and a lower risk of death compared to internal fixation. While the preliminary data supporting the use of arthroplasty for minimally displaced fractures is promising, the necessary evidence to make this significant practice change remains lacking.

The eventual definitive trial has significant potential to change clinical practice and optimize patient outcomes for individuals that experience a minimally displaced FNF. Treating minimally displaced FNFs with arthroplasty, instead of internal fixation, would be a paradigm shift in clinical care. This pilot study will demonstrate feasibility of the definitive trial and be used to refine aspects of the study protocol as necessary. If feasibility is successfully demonstrated, the pilot activities will be considered a vanguard phase for the definitive clinical trial.

Adult patients ages 60 years or older with a low-energy minimally displaced femoral neck fracture treated with surgery will be eligible to participate in the study. Patients will be randomized to receive either hip arthroplasty or internal fixation. Patients will be followed for 1 year, with visits occurring at 6 weeks, 4 months, 8 months, and 1 year after fracture. At each follow-up, mortality, ambulation, days at home, and health status will be collected.

The primary objective is to assess feasibility of the trial and to collect information to inform the design of the definitive trial. The feasibility outcomes will include participant enrollment, adherence to treatment allocation, data collection methods, and compliance with key aspects of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years of age or older.
* Complete fracture of the femoral neck (AO/OTA 31B) confirmed with anteroposterior and lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Minimally displaced fracture that could be, in the judgment of the attending surgeon, optimally managed with either arthroplasty or in situ internal fixation without reduction.
* Low energy injury mechanism defined as a fall from standing height.
* Informed consent obtained from patient or proxy.
* Surgeons with expertise in total hip arthroplasty, hemiarthroplasty, and internal fixation are available to perform surgery. Note: Surgeons do not need to be experts in all techniques.

Exclusion Criteria:

* Unable to ambulate 10 feet pre-injury with any assistance.
* Associated lower extremity injury that prevents post-operative weightbearing.
* Retained hardware around the hip that precludes either study treatment.
* Infection around the hip (soft tissue or bone).
* Pathologic fracture with a lytic lesion in the femoral neck that precludes internal fixation.
* Patient is too ill, in the judgement of the attending surgeon, for internal fixation.
* Patient is too ill, in the judgement of the attending surgeon, for arthroplasty.
* Unable to obtain informed consent due to language barriers.
* Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
* Currently enrolled in a study that does not permit co-enrollment.
* Prior enrollment in the trial.
* Other reason to exclude the patient, as approved by the Methods Centre.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Participant Enrollment | 12 months
  Participant enrollment will be assessed by monitoring screening and enrollment metrics, including:
  * Proportion of clinical sites initiated and able to screen consecutive patients with minimally displaced FNF
  * Proportion of patients who are screened for eligibility to participate in the trial
  * Proportion of patients who meet the eligibility criteria
  * Proportion of patients who provide informed consent
  * Proportion of time required to enroll at least four participants per clinical site
  * Proportion of reasons for exclusion.
Feasibility of Treatment Allocation | 12 months
  Feasibility of the treatment allocation will be assessed using the following metrics:
  * Adherence to arthroplasty treatment allocation
  * Adherence to internal fixation treatment allocation
Refine Data Collection Methods | 12 months
  To refine the data collection methods, the following metrics will be reviewed:
  * Proportion of participants with missing data
  * Review of missing data to identify data fields that are not feasible to collect
  * Data errors to identify ways to improve the flow of the case report forms (CRFs) and data collection
Assess Protocol Compliance | 12 months
  The following metrics will be used to assess compliance with the protocol:
  * Proportion of randomization errors
  * Proportion of participants who complete each follow-up visit
  * Proportion of participants who withdraw from the trial (withdrawal of consent)
  * Proportion of participants who cannot be located (loss to follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Slobogean, MD, Principal Investigator — University of Maryland, Baltimore; Sheila Sprague, PhD, Principal Investigator — McMaster University; Joseph Patterson, MD, Principal Investigator — University of Southern California
Locations (12):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Capital Region Health, Largo, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
- Vall d'Hebron University Hospital, Barcelona, Spain